CLINICAL TRIAL: NCT00000811
Title: A Randomized, Phase II/III, Double-Blind, Two-Armed Study of Micronized Atovaquone and Azithromycin (AT/AZ) as Compared to Trimethoprim-Sulfamethoxazole (TMP/SMX) in the Prevention of Serious Bacterial Infections When Used in Children Aged 3 Months to 19 Years With HIV Infection
Brief Title: A Study to Compare Different Drugs Used to Prevent Serious Bacterial Infections in HIV-Positive Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Pfizer (Industry); Glaxo Wellcome (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 254; PACTG 254; 11231 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Bacterial Infections; Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents; AIDS-Related Complex; Azithromycin; Bacterial Infections; atovaquone
MeSH Terms: conditions — Bacterial Infections; Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Azithromycin; Atovaquone; Trimethoprim, Sulfamethoxazole Drug Combination

INTERVENTIONS:
Drug: Azithromycin
Drug: Atovaquone
Drug: Sulfamethoxazole-Trimethoprim

SUMMARY:
This study compares 2 different treatments administered to try to prevent serious bacterial infections (such as pneumonia) in HIV-positive children. A combination of drugs (azithromycin plus atovaquone) will be compared to sulfamethoxazole-trimethoprim (SMX/TMP) alone. This study also evaluates the long-term safety and tolerance of these different drugs.

SMX/TMP is a commonly prescribed drug for the prevention of bacterial infections. However, the combination of azithromycin and atovaquone may be safer and more effective than SMX/TMP. This study compares the 2 treatments.

DETAILED DESCRIPTION:
Although SMX/TMP remains the drug of choice for PCP prophylaxis, drug sensitivity may limit its use. Atovaquone has demonstrated greater safety than SMX/TMP and thus is suitable as a candidate drug for treatment and prophylaxis of PCP. Azithromycin, with a broad anti-microbial spectrum (including mycoplasma and atypical mycoplasma), is an attractive prophylactic agent for use in children with HIV infection, due to its relative safety and once-daily dosing regimen. Therefore, the combination of atovaquone and azithromycin may offer broader antimicrobial coverage and greater safety than SMX/TMP.

Patients are randomized to receive either SMX/TMP or combination micronized atovaquone/azithromycin. Crossover to the alternative regimen may occur if serious toxicity is observed. Patients are monitored for occurrence of serious bacterial infections or PCP breakthrough, and when a serious bacterial infection occurs, patients are crossed over to the alternative regimen. Treatment continues until 2 years after the last patient is enrolled. The first 30 patients will undergo a pharmacokinetic profile. Patients are followed every 4 weeks for the first 4 months, then every 8 weeks thereafter. [AS PER AMENDMENT 05/28/99: This study was closed to infants and children age 19 months and older on 2/15/99; the study is now open to infants age 3 to 18 months (Stage II). Patients who are age 24 months or older at the time of Stage I closure will have end-of-study evaluations and will no longer be followed on protocol. Patients who are less than 24 months of age at the time of Stage I closure will be allowed to continue in the current version of the protocol. Enrollment for children age 3 to 18 months will continue until 50 subjects have been randomized. Because Stage II is an unblinded study, patients who are less than 24 months of age currently enrolled on Version 4.0 will have their study medication regimen unblinded and their atovaquone dose increased.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive.
* Are between the age of 3 months and 18 months (consent of parent or guardian required). (This study has been changed. In an earlier version, patients up to 19 years old were eligible.)
* Are at risk for developing pneumonia and need preventive treatment.
* Have a CD4 count of less than 1,500 cells/mm3 if under 1 year of age or a CD4 count of less then 500 cells/mm3 if between 1 and 2 years of age.

Exclusion Criteria

Children will not be eligible for this study if they:

* Have an infection that requires treatment.
* Are allergic to atovaquone, azithromycin, or SMX/TMP.
* Have serious diarrhea for more than 1 week.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 690
Dates: Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne M Dankner, Study Chair; Ram Yogev, Study Chair; Walter T Hughes, Study Chair
Locations (75):
- United States (72):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Earl K Long Early Intervention Clinic, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Cooper Hosp - Univ Med Ctr / UMDNJ - New Jersey Med Schl, Camden, New Jersey
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - Children's Hosp Pact Prog / Children's Hosp of Buffalo, Buffalo, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Ngo LY, Yogev R, Dankner WM, Hughes WT, Xu J, Unadkat J. Pharmacokinetics of azithromycin (AZ) when administered alone and with atovaquone (AT). Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:174 (abstract no 506)
- [Background] Ngo LY, Yogev R, Dankner WM, Hughes WT, Burchett S, Xu J, Sadler B, Unadkat JD. Pharmacokinetics of azithromycin administered alone and with atovaquone in human immunodeficiency virus-infected children. The ACTG 254 Team. Antimicrob Agents Chemother. 1999 Jun;43(6):1516-9. doi: 10.1128/AAC.43.6.1516. PMID 10348786
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891